CLINICAL TRIAL: NCT04869007
Title: The Impact of Cesarean Scar Defects on the Success of Assisted Human Reproduction: The Prospective NICHE-ART Study
Brief Title: The Impact of Cesarean Scar Defects on the Success of Assisted Human Reproduction
Acronym: NICHE-ART
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC20_0156
Record Dates: First submitted 2020-08-16; First posted 2021-05-03 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Cesarean Section; Dehiscence
Keywords: ceasarean scar defect; Isthmocele; in vitro Fecondation; Clinical pregnancy; live birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with a history of cesarean section and a hysterosonographically diagnosed isthmocoele: For patients who agreed to participate in the study, a specific measurement is made during the hysterosonography examination in order to determine the presence or absence of an isthmocele. Inclusion in the study is validated after a successful hysterosonography examination that confirms the presence or absence of an isthmocele. The patients are then attributed either to the: "isthmocele +" group or "isthmocele -" group.
  Interventions: Device: hysterosonography
- Patients with a history of cesarean section without isthmocoele hysterosonographically diagnosed: For patients who agreed to participate in the study, a specific measurement is made during the hysterosonography examination in order to determine the presence or absence of an isthmocele. Inclusion in the study is validated after a successful hysterosonography examination that confirms the presence or absence of an isthmocele. The patients are then attributed either to the: "isthmocele +" group or "isthmocele -" group.
  Interventions: Device: hysterosonography

INTERVENTIONS:
Device: hysterosonography — Isthmocele mesured by hysterosonography before ART procedure

SUMMARY:
The prevalence of Caesarean sections continues to increase around the world. In France, the proportion of Caesarean sections has doubled from 11% in 1981 to 20,2% in 2016, bringing with it an increase in the risk of obstetrical complications.

Uterine defects, or Isthomcele, first defined by Morris in 1995 as a scarring abnormality with a dehiscence of the hysterotomy following a caesarean section. This purely iatrogenic pathology can cause inter-menstrual bleeding or pelvic pain.

Several definitions of isthmosceles exist in scientific literature with variations according to the nature of the reference examination chosen and the measurements made. However, for the majority of authors, isthmoceles are characterized by a residual myometrial thickness of less than 3 millimetres in the sagittal plane. The prevalence of isthmoceles amoung patients with a unicicatricial uterus is about 61%.

Currently, the main diagnostic technique for isthmoceles are 2D or 3D ultrasound and hysterosonography.

Small, non-controlled studies have found that surgical treatment of the isthmocele is effective in reducing metrorrhagia. In these studies, the authors noted that patients with metrorrhagia were also more frequently affected by secondary infertility.

A small number of non-comparative studies with a low level of evidence have looked into the efficacy of surgical treatment of isthmoceles on related symptoms: metrorraghia, pelvic pain and/or secondary infertility. Their results show an idiopathic secondary infertility rate in the presence of isthmoceles prior to surgical treatment of approximately 66%. Significantly higher pregnancy rates after treatment suggest that the surgical management of isthmoceles is worthwhile. However, these data suffer from not negligible selection bias.

The initial findings concerning fertility after surgical repair seem promising and some teams propose systematic surgical management of the isthmocele before a technique of assisted reproduction (ART) although without any evidence in literature.

Isthmocele surgery can result in uterine perforations, adhesions and intrauterine synechia known to be detrimental to future fertility.

The efficacy of surgical management of surgey must therefore be demonstrated prior to any attempts at treatment. This will require large prospective studies based on a consensual definition of isthmocele. The diagnosis using Hysterosonography is currently considered as the "gold standard" examination.

The main hypothesis of our study is that a significant isthmocele, defined by a residual myometrial thickness of less than 3mm, measured in the sagittal plane by hysterosonography, could alter the results of ART.

DETAILED DESCRIPTION:
The study has a multicentric, parallel group, comparative, non-interventional, exploratory and prospective design.

Definition of isthmocele: defined as a dehiscence of the hysterotomy following a caesarean section. The residual myometrial thickness is less than 3mm, measured in the sagittal plane by hysterosonography.

The presence or absence of an isthmocele according to this definition will allow for the distribution of patients into one of two study groups : "isthmocele +" or "isthmocele -".

Definition of clinical pregnancy rate: defined as the presence of an intrauterine gestational sac and an embryo with cardiac activity visualized during an ultrasound examination at 7 weeks after embryo transfer.

Methods : During the initial ART consultation, the study is presented (oral information and distribution of a brochure) to patients consulting for infertility and with a history of cesarean section. It is during this consultation that the ART treatment assessment (blood tests and imaging: ultrasound and hysterosonography) is prescribed. If they agree to take part in the study, the non-opposition of eligible patients is collected during this consultation (pre-inclusion). Furthermore, among patients who agreed to participate in the study, socio-demographic data and the couple's medical history are collected during this initial consultation.

For patients who agreed to participate in the study, a specific measurement is made during the hysterosonography examination in order to determine the presence or absence of an isthmocele. Inclusion in the study is validated after a successful hysterosonography examination that confirms the presence or absence of an isthmocele. The patients are then attributed either to the: "isthmocele +" group or "isthmocele -" group.

During the second ART consultation, the results of the treatment assessment are collected, in particular the presence or absence of an isthmocele on the hysterosonography examination.

Subsequently, the data relative to ovarian stimulation, the methods of triggering and embryo transfer are collected prospectively by the investigator or co-investigators.

As part of the standard ART treatment, blood HCG tests are carried out 14 days after embryo transfer in order to detect a possible pregnancy. If the blood HCG levels are positive, the test is repeated 48 hours later and again a week later to survey the evolution of the blood HCG levels. At 6 to 7 weeks after oocyte puncture, an ultrasound scan is performed in the ART department if the blood HCGs level is greater than 10 IU/L with a satisfactory evolution after 48 hours. This data is collected for research purposes.

In the case of pregnancy and delivery in the same hospital as the ART treatment, obstetrical data is collected by the investigators or co-investigators from the obstetrical file. In the case of delivery at another facility, patients were contacted by telephone one year after a positive pregnancy test (HCG).

Discussion: No individual benefit is expected from this study since the management of the patients included corresponds to standard practice.

Concerning the collective benefits, if the conclusions of this study allow for the confirmation of our hypothesis (reduction in the pregnancy rate in the presence of a significant isthmocele), this could lead to a change in clinical practices in patients treated with ART. Indeed, surgical management of the isthmocele could be discussed prior to ART by informing the patient of the benefit-risk balance of the operation.

If our hypothesis of reduced fertility in the presence of isthmoceles is confirmed, further studies should ideally be carried out in order to demonstrate that the surgical management of isthmoceles improves the results of ART before systematically offering surgery to patients.

Trial Registration : The research protocole has been approuved by the relevant French authorities Comité de Protection des Personnes Sud Méditerranée IV on the 10th of November 2020 and recorded prospectively (before the inscription of the first participant) under the number ID-RCB : 2020-A02068-31.

ELIGIBILITY:
Inclusion criteria :

* Patients with a history of at least one cesarean section (single or multi-scarred uterus).
* Age between 18 and 43 years old
* Secondary infertility requiring ART techniques (FIV or FIV ICSI).
* A Hysterosonography examination as part of the pre-ART assessment allowing for the detection of the presence of an isthmocele.
* French speaking patients
* Patient affiliated to or beneficiary of a social security scheme

Non-inclusion criteria :

- Refusal to participate in the study.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients referred to an ART procedure for secundary infertility with a history of at least one cesarean section (single or multi-scarred uterus).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Significant isthmocele and clinical pregnancy rates after ART procedure | 12 months
  A significant isthmocele (defined by a residual myometrial thickness of less than 3 mm in the sagittal plane, mesured by hysterosonography) could alter the results of ART (pregnancy rates). Definition of clinical pregnancy rate: defined as the presence of an intrauterine gestational sac and an embryo with cardiac activity visualized during an ultrasound examination at 7 weeks after embryo transfer

SECONDARY OUTCOMES:
The secondary objectives of the study explore the associations between the presence of an isthmocele and other criteria evaluating the results of IVF in patients with a scarred uterus | 12 months
  The secondary objectives of the study explore the associations between the presence of an isthmocele and other criteria evaluating the results of IVF (IVF or IVF ICSI) in patients with a scarred uterus (single or multi-scarred)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LEGENDRE, MD PhD, Principal Investigator — UH Angers
Locations (9):
- France (9):
  - UH Angers, Angers
  - University Hospital of Brest, Brest
  - Hospital Center Sud Francilien, Corbeil-Essonnes
  - Creteil University Hospital, Créteil
  - University Hospital of Nimes, Nîmes
  - Tenon Hospital Paris, Paris
  - La Sagesse Clinic, Rennes
  - University Hospital of Rennes, Rennes
  - University Hospital of Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Spiezio Sardo A, Di Carlo C, Minozzi S, Spinelli M, Pistotti V, Alviggi C, De Placido G, Nappi C, Bifulco G. Efficacy of hysteroscopy in improving reproductive outcomes of infertile couples: a systematic review and meta-analysis. Hum Reprod Update. 2016 Jun;22(4):479-96. doi: 10.1093/humupd/dmw008. Epub 2016 Mar 23. PMID 27008893
- [Background] Bij de Vaate AJ, van der Voet LF, Naji O, Witmer M, Veersema S, Brolmann HA, Bourne T, Huirne JA. Prevalence, potential risk factors for development and symptoms related to the presence of uterine niches following Cesarean section: systematic review. Ultrasound Obstet Gynecol. 2014 Apr;43(4):372-82. doi: 10.1002/uog.13199. PMID 23996650
- [Background] Donnez O, Jadoul P, Squifflet J, Donnez J. Laparoscopic repair of wide and deep uterine scar dehiscence after cesarean section. Fertil Steril. 2008 Apr;89(4):974-80. doi: 10.1016/j.fertnstert.2007.04.024. Epub 2007 Jul 10. PMID 17624346
- [Background] Osser OV, Jokubkiene L, Valentin L. High prevalence of defects in Cesarean section scars at transvaginal ultrasound examination. Ultrasound Obstet Gynecol. 2009 Jul;34(1):90-7. doi: 10.1002/uog.6395. PMID 19499514
- [Background] Jeremy B, Bonneau C, Guillo E, Paniel BJ, Le Tohic A, Haddad B, Madelenat P. [Uterine ishtmique transmural hernia: results of its repair on symptoms and fertility]. Gynecol Obstet Fertil. 2013 Oct;41(10):588-96. doi: 10.1016/j.gyobfe.2013.08.005. Epub 2013 Oct 4. French. PMID 24094595
- [Derived] Astruc A, Deseine D, Spiers A, Boguenet M, May-Panloup P, Bouet PE, Legendre G. Impact of caesarean scar defects on the success of assisted human reproduction: the NICHE-ART prospective French cohort study protocol. BMJ Open. 2024 Dec 7;14(12):e092011. doi: 10.1136/bmjopen-2024-092011. PMID 39645254